CLINICAL TRIAL: NCT05107102
Title: Value of Myocardial Work for Prediction of Left Ventricular Remodeling in Patients With ST-Elevation Myocardial Infarction Treated by Primary Percutaneous Intervention
Brief Title: Myocardial Work for Prediction of Left Ventricular Remodeling in Patients With STEMI
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: STEMI-myocardial work
Record Dates: First submitted 2021-10-24; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: ST-Segment Elevated Myocardial Infarction
Keywords: ST-segment elevated myocardial infarction; myocardial work; left ventricular remodeling
MeSH Terms: conditions — Ventricular Remodeling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with LVR(left ventricular remodeling)
- patients without LVR(left ventricular remodeling)

SUMMARY:
The study intends to investigate the alteration of regional myocardial work in patients with acute anterior myocardial infarction underwent primary percutaneous coronary intervention (PCI), and compare the distribution of regional myocardial work in patients with/without early remodeling at acute phase and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Anterior myocardial infarct (anterior myocardial infarct is defined as persistent chest pain for 30 mins at least, with ST-segment elevation of at least 0.2 mV in two or more contiguous precordial leads) within 12 hours after onsets of symptom;
* Left anterior descending (LAD) as culprit vessel, with TIMI 0-1 grade.

Exclusion Criteria:

* significant valvular disease;
* cardiomyopathy; l
* left bundle branch block;
* atrial fibrillation;
* previous myocardial infarction (MI);
* history of cardiac surgery;
* pacemaker implantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anterior STEMI who underwent primary PCI <12 hours after symptom onset were consecutive enrolled in our center.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Delta-work efficiency by echocardiography | 24-72 hours after PCI
  A novel tool for non-invasive myocardial work(MW) assessment has been introduced to evaluate myocardial performance.MW was calculated as a function of time through a combination of LV global longitudinal strain(GLS) data and an estimated LV pressure curves. Work efficiency (WE) was calculated from the ratio of the constructive work to the sum of constructive and wasted work, expressed as a percentage.The values of culprit regional WE was expressed as WE-LAD.The values of non-culprit regional WE was expressed as WE-nonLAD.The absolute differences of the WE was calculated as the values of non-culprit regional WE minus the values of culprit regional WE, and noted as delta-WE.

SECONDARY OUTCOMES:
Global work index by echocardiography | 24-72 hours, 3-month after PCI
  Global work index (GWI) is classified as total work within the area of the LV pressure-strain loop calculated from mitral valve closure to mitral valve opening.
Global constructive work by echocardiography | 24-72 hours, 3-month after PCI
  Global constructive work (GCW) was defined as work contributing to LV ejection performed during shortening in systole and work performed during lengthening in isovolumic relaxation.
Global work efficiency by echocardiography | 24-72 hours, 3-month after PCI
  Global work efficiency (GWE) was calculated from the ratio of the constructive work to the sum of constructive and wasted work, expressed as a percentage.
Work index-LAD | 24-72 hours, 3-month after PCI
  Work index in left anterior descending(LAD) territory.
Constructive work-LAD | 24-72 hours, 3-month after PCI
  constructive work in left anterior descending(LAD) territory.
Work efficiency-LAD | 24-72 hours, 3-month after PCI
  Work efficiency in left anterior descending(LAD) territory.

CONTACTS AND LOCATIONS:
Overall Officials: Song Ding, MD,PHD, Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang W, Zhao H, Wan F, Shen XD, Ding S, Pu J. Inhomogeneous Distribution of Regional Myocardial Work Efficiency Predicts Early Left Ventricular Remodeling After Acute Anterior Myocardial Infarction Treated With Primary Percutaneous Intervention. Front Cardiovasc Med. 2022 Jul 27;9:922567. doi: 10.3389/fcvm.2022.922567. eCollection 2022. PMID 35966524